CLINICAL TRIAL: NCT01118754
Title: Phase I/II Prospective, Randomized, Double Masked, Parallel-Group, Multi-centered Study Assessing the Safety and Efficacy of Two Concentrations of DE-101 Compared to Placebo for the Treatment of Dry Eye Disease
Brief Title: Study Assessing Safety and Efficacy of DE-101 Ophthalmic Suspension in Dry Eye Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26-004
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Dry Eye
Keywords: Santen; Dry; Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DE-101 ophthalmic suspension high dose (Experimental)
  Interventions: Drug: DE-101 ophthalmic suspension
- DE-101 ophthalmic suspension low dose (Experimental)
  Interventions: Drug: DE-101 ophthalmic suspension
- DE-101 ophthalmic suspension vehicle (Placebo Comparator)
  Interventions: Drug: DE-101 ophthalmic suspension; Drug: DE-101 ophthalmic suspension vehicle

INTERVENTIONS:
Drug: DE-101 ophthalmic suspension — Ophthalmic suspention; QID
Drug: DE-101 ophthalmic suspension — Ophthalmic suspension; QID
  Arms: DE-101 ophthalmic suspension low dose
Drug: DE-101 ophthalmic suspension vehicle — ophthalmic suspension vehicle; QID
  Arms: DE-101 ophthalmic suspension vehicle

SUMMARY:
The purpose of this study is to evaluate if DE-101 ophthalmic suspension will safely and effectively improve signs and or symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of dry eye defined by protocol
* 18 years or older, and sign written informed consent
* negative pregnancy test and utilizing reliable contraceptive throughout study

Exclusion Criteria:

* use of any topical ocular medications
* any ocular surgery within 90 days of study
* laser refractive surgery within one year of study
* ocular, lid disease/abnormalities that may interfere with the study
* corneal transplants
* uncontrolled systemic conditions
* females who are pregnant or nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception
* participated in another drug trial within 30 days prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Total fluorescein corneal staining | 8 weeks
Ocular Symptom Severity | 8 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Inglewood, California
  - Torrance, California
  - Bloomfield, Connecticut
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Gretna, Louisiana
  - Bangor, Maine
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - San Antonio, Texas